CLINICAL TRIAL: NCT07138911
Title: Effect of Home-based Exercise Plan Mediated by Use of Digital Health App on Kinesiophobia and Functional Capacity in Sedentary Post Myocardial Infarction Patient.
Brief Title: Effect of Home-based Exercise Plan Mediated by Use of Digital Health App on Kinesiophobia and Functional Capacity
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Noureen Begum
Record Dates: First submitted 2025-08-18; First posted 2025-08-24 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Myocardial Infarction; Kinesiophobia; Sedentary Behavior
Keywords: Digital health app; Functional capacity; Kinesiophobia; Myocardial Infarction; Sedentary
MeSH Terms: conditions — Myocardial Infarction; Kinesiophobia; Sedentary Behavior | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Home based exercise plan mediated by use of mobile health app
  Interventions: Other: Intervention group
- Control Group (Active Comparator): Home based exercise plan
  Interventions: Other: Control group

INTERVENTIONS:
Other: Intervention group — Walking at home for 15-30 minutes 3 times per day for 4 weeks. Activity plan is calendar on mobile health app. Mobile placed in pocket or bag before starting walk and mark activity on calendar.
  Arms: Intervention group
Other: Control group — Walking at home for 15-30 minutes 3 times per day for 4 weeks. Manual record of walking and date.
  Arms: Control Group

SUMMARY:
To evaluate the effect of home-based exercise plan mediated by a digital health application on kinesiophobia and functional capacity in sedentary post myocardial infarction patients. Evidence suggest that digital health application significantly improve physical activity level in patient following cardiac event by providing personalized exercise plan, real time feed back, progress tracking and motivational features which enhanced adherence and engagement in rehabilitation program. This study could offer a viable le solution for overcoming barrier to rehabilitation particularly for those unable to access traditional clinic-based program

DETAILED DESCRIPTION:
Mobile health (m health) strategies to increase adherence to physical activity is a promising approach. Mobile technology has become more integrated with health care and use of mobile health apps has become feasible for even the most novice users. Mobile health app can be effective adjuncts for the management of chronic condition and have a positive impact on long term behavior. The mobile health app promote the physical activity maintenance after cardiac rehabilitation. Recently, researchers have stated that mobile health intervention promoting the physical activity in the patient of cardiovascular disease. Mobile health intervention promote physical activity and daily step count after completing cardiac rehab.

ELIGIBILITY:
Inclusion Criteria:

* 3 months post myocardial infarction patient
* Sitting hours >8
* IPAQ < 600 Mets minutes

Exclusion Criteria:

* Unstable Angina
* Recurrent Myocardial infarction
* Recent surgery or Procedure
* Heart failure, Arrhythmia

Ages: 30 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 88 (Estimated)
Dates: Start 2025-08-13 (Estimated); Primary Completion 2026-01-15 (Estimated); Study Completion 2026-02-15 (Estimated)

PRIMARY OUTCOMES:
Kinesiophobia | 4 Weeks
  Changes from baseline to 4 weeks after intervention, measured through the TSK-SV Heart specifically focuses on assessing Kinesiophobia in the context of cardiac conditions or symptoms. It include questions related to fear of engaging in physical activity due to concerns about cardiac events (such as heart palpitations, chest pain, or shortness of breath) during exercise or daily activities. The 17 item TSK total scores range from 17 to 68 where the lowest 17 means no or negligible Kinesiophobia, and the higher scores indicate an increasing degree of Kinesiophobia.
Functional Capacity | 4 Weeks
  Changes from baseline to 4 weeks after intervention, measured through six minute walk test which is a sub-maximal exercise test used to assess functional capacity and endurance. The distance covered over a time of 6 minutes is used as the outcome by which to compare changes in performance capacity.

CONTACTS AND LOCATIONS:
Overall Officials: Mehwish Waseem, MS-CPPT PhD*, Principal Investigator — Riphah International University
Locations (1):
- Polyclinic Hospital, Islamabad, Federal, Pakistan

IPD SHARING:
Plan to Share IPD: No